CLINICAL TRIAL: NCT00555568
Title: Mechanisms of Action and Outcome in Peer Support Groups
Brief Title: Mechanisms of Action and Outcome
Acronym: Peer Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D4464-R
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Mental Disorders
Keywords: mental health; group processes
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Peer-led Groups (Experimental): Arm 1 is a 3-month recovery-focused mental health education and support group led by peer facilitators
  Interventions: Behavioral: recovery oriented mental health peer support group
- Clinician-led Groups (Experimental): Arm 2 is a 3-month recovery-focused mental health education and support group led by a mental health clinician
  Interventions: Behavioral: recovery-oriented mental health clinician-led group
- Treatment as Usual (No Intervention): Arm 3 is treatment as usual (no intervention)

INTERVENTIONS:
Behavioral: recovery oriented mental health peer support group — This is a recovery-focused mental health education and support group led by peer facilitators
  Arms: Peer-led Groups
Behavioral: recovery-oriented mental health clinician-led group — This is a recovery-focused mental health education and support group led by a mental health clinician
  Arms: Clinician-led Groups

SUMMARY:
The objective of this study is to examine the mechanisms of action and outcome in mental health peer support groups. The study design is a randomized trial in which participants are assigned to one of three study arms: a recovery oriented mental health group led by peer facilitators (Vet-to-Vet), a recovery oriented group led by a clinician, or "treatment as usual." Qualitative and quantitative methods will be used to assess substantive content and process of the recovery groups, as well as mental health and recovery outcomes.

DETAILED DESCRIPTION:
Background: Rehabilitation and recovery services for individuals with psychiatric disorders are an important focus of the Veterans Health Administration. In FY 2004, 847,131 veterans (17.4% of VHA patients) received specialized VHA mental health services at a cost of almost $2 billion. In June 2004, Secretary Principi initiated a Mental Health Task Force to improve mental health care for veterans. The resulting comprehensive strategic plan, A Road Map for Transforming VA Mental Health Care" presented two central recommendations: 1) emphasize the recovery model at every medical center, and 2) develop and implement the full continuum of recovery-oriented mental health services. A recovery oriented mental health system is one that fosters self-determination, hope, and empowerment. Peer/consumer support groups, which provide a forum for mutual acceptance, empowerment, information, education, advocacy, skills training, and community reintegration are an important component of this plan, and have been implemented in a number of VHA centers.

Objectives: The objectives of the proposed research are to assess the content and impact of VHA mental health peer support groups for recovery from mental illness. Specifically, we will: a) examine the structure, process and outcome of two models of recovery-oriented group treatment for mental health-peer/consumer support groups led by peer facilitators (Vet-to-Vet program), and recovery-oriented groups led by a clinician; b) assess and compare empowerment, social support, traditional outcomes (psychiatric and substance abuse symptoms, community functioning) and recovery-oriented outcomes (hope, strength/resiliency) in each type of program; and c) test a model in which recovery-oriented outcomes are mediated by empowerment and social support.

Methods: The study will use a research design in which participants are randomly assigned to attend an existing peer facilitator-led support group, a clinician-led recovery-oriented group, or "treatment as usual". The sample will include 300 individuals receiving outpatient mental health services at one of two VA sites: Bedford, MA or West Haven, CT. Qualitative and quantitative methods will be used to address the research objectives. We will observe and tape record a sample of group meetings, and interview participants and group leaders (consumer-facilitators or clinicians) to analyze and understand the "ingredients" (structure and content) of these groups. We will use standardized measures of self-efficacy, empowerment and social support to determine effects of group type on participants' feelings of empowerment and social support, and whether empowerment and social support result in better outcomes. We will assess recovery-oriented (hope, optimism, strength and resilience) and traditional (symptom and functioning) outcomes. Qualitative data from group observations and interviews will be used to explore what other factors might explain the effects of participation in peer-support and clinician-led groups. Quantitative measures will be analyzed using regression modeling in an "intent to treat" approach. Path analysis that entails a series of regression models will be used to test the hypothesized mediation effect.

Significance to VA: The VA has made a clear commitment to implementation of peer-support programs as part of a recovery-oriented transformation of its mental health service system. However, there is currently no published research reporting the processes or outcomes of these programs. This study will provide valuable information regarding if, why and how peer support groups, as well as clinician-led recovery-oriented groups, benefit veterans with mental illness. This information will be valuable in guiding implementation of such programs across the country.

ELIGIBILITY:
Inclusion Criteria:

* veteran in treatment for a psychiatric disorder at a participating study site

Exclusion Criteria:

* currently participating in a recovery group that constitutes an intervention arm of this research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan V. Eisen, PhD BA, Principal Investigator — VA New England Health Care System; Jack A Clark, PhD, Principal Investigator — VA New England Health Care System
Locations (2):
- United States (2):
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA New England Health Care System, Bedford, Massachusetts

REFERENCES:
- [Result] Eisen SV, Schultz MR, Mueller LN, Degenhart C, Clark JA, Resnick SG, Christiansen CL, Armstrong M, Bottonari KA, Rosenheck RA, Sadow D. Outcome of a randomized study of a mental health peer education and support group in the VA. Psychiatr Serv. 2012 Dec;63(12):1243-6. doi: 10.1176/appi.ps.201100348. PMID 23203360
- [Result] Beehler S, Clark JA, Eisen SV. Participant experiences in peer- and clinician-facilitated mental health recovery groups for veterans. Psychiatr Rehabil J. 2014 Mar;37(1):43-50. doi: 10.1037/prj0000048. PMID 24660950
- [Result] Bottonari KA, Schultz MR, Resnick SG, Mueller L, Clark J, Sadow DC, Eisen SV. Peer-led vs. Clinician-led Recovery-Oriented Groups: What Predicts Attendance by Veterans? International Journal of Psychosocial Rehabilitation. 2012 Jan 1; 16(2):96-113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three cohorts of veterans were recruited from each of two sites. Those assigned to a peer-led group participated in the Vet-to-Vet program. Those assigned to a clinician-led group participated in a recovery-oriented group led by a clinician. Those assigned to 'treatment-as-usual' continued with their usual treatment.
Groups:
- Arm 1: Peer-led Group: Arm 1 is a 3-month recovery-focused mental health education and support group led by peer facilitators
- Arm 2: Clinician Led Group: Arm 2 is a 3-month recovery-focused mental health education and support group led by a mental health clinician
- Arm 3: Treatment as Usual: Arm 3 is treatment as usual (no intervention)
Period: Overall Study
Arm/Group | Arm 1: Peer-led Group | Arm 2: Clinician Led Group | Arm 3: Treatment as Usual
Started | 100 | 98 | 100
Completed | 74 | 82 | 84
Not Completed | 26 | 16 | 16
Not completed — Lost to Follow-up | 26 | 16 | 16

BASELINE CHARACTERISTICS:
Population: veterans treated for a mental health condition at one of 2 VA medical centers
Groups:
- Arm 1: Peer-Led Group: Arm 1 is a 3-month recovery-focused mental health education and support group led by peer facilitators
  recovery oriented mental health peer support group: This is a recovery-focused mental health education and support group led by peer facilitators
- Arm 2: Clinician-Led Group: Arm 2 is a 3-month recovery-focused mental health education and support group led by a mental health clinician
  recovery-oriented mental health clinician-led group: This is a recovery-focused mental health education and support group led by a mental health clinician
- Total: Total of all reporting groups
Arm/Group | Arm 1: Peer-Led Group | Arm 2: Clinician-Led Group | Arm 3: Treatment as Usual | Total
Number analyzed (Participants) | 100 | 98 | 100 | 298
Age, Customized [Number; unit: participants]
  < 35 years | 7 | 8 | 3 | 18
  35-50 years | 31 | 38 | 24 | 93
  51-60 years | 44 | 36 | 52 | 132
  >60 years | 18 | 16 | 21 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 7 | 22
  Male | 95 | 88 | 93 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 8 | 28
  Not Hispanic or Latino | 88 | 90 | 92 | 270
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 22 | 32 | 23 | 77
  White | 66 | 58 | 66 | 190
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 8 | 11 | 31
Region of Enrollment [Number; unit: participants]
  United States | 100 | 98 | 100 | 298

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation
Description: Patient activation refers to patient knowledge skill and confidence for self-management.
  Full name of the scale is Patient Activation Measure (PAM). Scale response options range from 1-4 and scores can range from 13-52. Higher values indicate greater activation. No subscales are used.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 2: Clinician-led Group: Arm 2 is a 3-month recovery-focused mental health education and support group led by a mental health clinician
Arm/Group | Arm 1: Peer-led Group | Arm 2: Clinician-led Group | Arm 3: Treatment as Usual
Number analyzed (Participants) | 74 | 82 | 84
units on a scale | 29.12 (5.91) | 28.82 (6.48) | 29.21 (5.80)

2. Primary Outcome: Empowerment
Description: Empowerment is measured by the "Making Decisions" instrument. Response options range from 1-4 and scores can range from 28-112. Higher scores indicate more empowerment.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Peer-led Group | Arm 2: Clinician-led Group | Arm 3: Treatment as Usual
Number analyzed (Participants) | 74 | 82 | 84
units on a scale | 80.20 (6.66) | 80.85 (8.00) | 81.15 (8.37)

3. Primary Outcome: Social Support
Description: Social Support was assessed by the Medical Outcomes Study Social Support Survey. Response options range from 1-5 and scores range from 19-95. Higher scores indicate greater social support
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Peer-led Group | Arm 2: Clinician-led Group | Arm 3: Treatment as Usual
Number analyzed (Participants) | 74 | 82 | 84
units on a scale | 63.18 (16.59) | 58.21 (19.00) | 64.30 (16.31)

4. Primary Outcome: VR-12 MCS
Description: VR-12 MCS refers to the Mental Health Component of the SF-12. The rating scale varies depending on the item. Scores range from 0-100; higher values indicate better mental health;
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Peer-led Group | Arm 2: Clinician-led Group | Arm 3: Treatment as Usual
Number analyzed (Participants) | 74 | 82 | 84
units on a scale | 47.16 (12.41) | 44.57 (13.30) | 47.18 (12.80)

5. Primary Outcome: Overall Mental Health (BASIS-24 Summary Score)
Description: BASIS-24 refers to the 24-item Behavior and Symptom Identification Scale. Responses range from 0-4; scores range from 0-4; higher values indicate greater symptom severity.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Peer-led Group | Arm 2: Clinician-led Group | Arm 3: Treatment as Usual
Number analyzed (Participants) | 74 | 82 | 84
units on a scale | 1.09 (0.65) | 1.24 (0.66) | 1.08 (0.65)

ADVERSE EVENTS:
Time Frame: from enrollment to completion of 3-month follow-up
Arm/Group | Arm 1: Peer-led Group | Arm 2: Clinician-led Group | Arm 3: Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/98 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/98 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes